CLINICAL TRIAL: NCT04065971
Title: Randomized, Placebo-controlled, Double-blind Study to Evaluate the Efficacy of 2LHERP® in Patients With Recurrent Orofacial Herpes Infections.
Brief Title: Randomized, Placebo-controlled, Double-blind Study of 2LHERP® in Orofacial Herpes Infections.
Acronym: HEARTH-OF
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Labo'Life (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LLB-2018-01
Record Dates: First submitted 2019-08-21; First posted 2019-08-22 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Herpes Simplex
MeSH Terms: conditions — Herpes Simplex

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2LHERP® arm (Experimental): Group N°1: 2LHERP® treatment (6 months of treatment)
  Interventions: Drug: 2LHERP®
- Placebo arm (Placebo Comparator): Group N°1: Placebo treatment (6 months of treatment)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 2LHERP® — The treatment schema consists in taking the content of one capsule a day, 15-30 minutes before breakfast, on an empty stomach, sequentially, according to capsules' numerical order: 1 through 10. When capsule number 10 is taken, capsule 1 of the next blister should be taken on the next day to continue the treatment. The duration of treatment will be 6 months of continuous intake of the content of 1 capsule/day.
  Other Names: 2LHERP
  Arms: 2LHERP® arm
Drug: Placebo — The treatment schema consists in taking the content of one capsule a day, 15-30 minutes before breakfast, on an empty stomach, sequentially, according to capsules' numerical order: 1 through 10. When capsule number 10 is taken, capsule 1 of the next blister should be taken on the next day to continue the treatment. The duration of treatment will be 6 months of continuous intake of the content of 1 capsule/day.
  Arms: Placebo arm

SUMMARY:
Herpes simplex virus (HSV) infection is very common, as most people will experience herpetic infection during their lifetime. The most common manifestation of HSV infection is sores which may appear at any age.

No specific antiviral therapy is available to totally cure herpetic infections and today, there is no treatment that allows the definitive eradication of the virus.

The 2LHERP® has been available for more than 20 years, and has received a marketing authorization in Belgium by the FAMHP. It is used as an immune regulator in the treatment of herpetic infections. Since 2LHERP® has been made available, clinical observational data collected on treated patients have shown the beneficial effect on the disappearance of herpetic recurrences.

The purpose of this placebo-controlled trial is to evaluate the efficacy of 2LHERP® on the treatment of herpetic infections in adults.

DETAILED DESCRIPTION:
The study duration will be 36 months with 24 months of inclusion (that may be extended if the expected number of patients is not reached after this period) and 12 months of follow-up.

Patients aged between 16 and 80 years who present recurrent orofacial herpes infections (6 or more episodes within the 12-months' period prior to their study entry).

The total number of patients to include will be 140 with 70 patients per group.

Primary objective:

Evaluation of the efficacy of 2LHERP® on the reduction of the number of recurrent orofacial herpes episodes at 12 months.

Secondary objectives:

Comparison of the efficacy of 2LHERP® vs placebo according to the following aspects:

1. number of episodes at 6 months,
2. time to first episode during the treatment,
3. duration of episodes,
4. symptomatology during the entire relapse time,
5. use of Rescue Medication (RM),
6. evaluation of impact on the quality of life,
7. safety issues.

Treatment phase:

* Group n°1 = 2LHERP® (6 months of treatment)
* Group n°2 = Placebo (6 months of treatment) Post-treatment follow-up phase: 6 months. Treatment will be considered successful if the number of herpetic episodes is reduced.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged 16-80 years,
* Patient presenting 6 or more episodes of orofacial herpes infections during the preceding 12-months' period (prior to the study entry),
* Woman of childbearing age under effective contraception,
* Patient reporting a current stable sexual relationship (steady sexual partner during study duration),
* Patient having faculties to understand and respect the constraints of the study,
* Signature of the Informed Consent Form.

Exclusion Criteria:

* Pregnant or breastfeeding woman,
* Patient under immunotherapy (including immunosuppressive treatment) or micro-immunotherapy received during last previous 6 months,
* Patient who had a suppressive antiviral therapy during last month,
* Patient who wishes to continue his/her suppressive antiviral therapy,
* Patient with known lactose intolerance,
* Patient who participated in a clinical study in the previous 3-month period,
* Patient who is not sufficiently motivated to engage in a follow-up period of 12 months, or likely to travel or to move before the end of the study,
* Patient with severe immunodeficiency disease requiring long term treatment (*) or under chemotherapy or radiotherapy or corticoid therapy,
* Patient under listed homeopathic or phytotherapy treatment,
* Patient using or addicted to recreational drugs.

(*) important renal or respiratory insufficiency, transplanted or grafted patients HIV/AIDS, terminal cancer.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2020-03-10 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the efficacy of 2LHERP® on the reduction of the number of recurrent orofacial herpes episodes at 12 months. | 12 months
  The primary objective of the study will be to evaluate the change from baseline within the number of episodes of herpes infections observed for 12 months, where the baseline value is the number of episodes experienced within the 12 months preceeding study enrolment.

SECONDARY OUTCOMES:
Remaining herpes infection recurrence free 12 months after treatment initiation (yes/no) | 12 months
  The objective of this outcome will be to compare the number of patients recurrence free for 12 months between the treated and the placebo group.
Remaining herpes infection recurrence free 6 months after treatment initiation (yes/no) | 6 months
  The objective of this outcome will be to compare the number of patients recurrence free for 6 months after treatment initiation between the treated and the placebo group.
Number of episodes of herpes infection observed at 6 months | 6 months
  The objective of this outcome will be to compare the number of herpetic episodes at 6 months and the baseline number of episodes.
Time to first recurrence of herpes infection during the treatment | 6 months
  The objective of this outcome will be to compare the time to first herpetic recurrence between the treated and the placebo group.
Mean duration of episodes, the duration for a given episode being defined as the number of days between the start of the episode and the last day before all symptoms recorded as 'none' for 2 consecutive days, in the patient diary | 12 months
  The objective of this outcome will be to compare the mean duration of the herpetic episodes between the treated and the placebo group.
Level of pain recorded daily as well as other associated symptomatology for orofacial pain, which will be consequently measured as area under the curve | 12 months
  The objective of this outcome will be to compare the level of pain during herpetic episodes between the treated and the placebo group.
Use of daily rescue medicine (RM), expressed with the cumulative number of days for the treatment period, the follow-up period and the entire study period | 12 months
  The objective of this outcome will be to compare the use of rescue medication during herpetic episodes between the treated and the placebo group.
Quality of life evaluated via a 6-items questionnaire | 6 and 12 months
  The objective of this outcome will be to compare the quality of life between the treated and the placebo group.
Occurrence of adverse events (AEs) and severe adverse events (SAEs), considered as related or not to the study drug | 6 months
  The objective of this outcome is to evaluate the safety of the treatment

CONTACTS AND LOCATIONS:
Locations (6):
- Belgium (6):
  - Private Practice, Beerzel
  - Cabinet privé, Beuzet
  - Clinique Saint-Luc (Bouge), Bouge
  - Private Practice, Linkebeek
  - Cabinet privé, Noirefontaine
  - Private Practice, Oisquercq

IPD SHARING:
Plan to Share IPD: No